CLINICAL TRIAL: NCT02036177
Title: A Prospective, Randomized, Single Blind, Two Arms Controlled Study to Confirm the Safety and Verify Performance of the IUB™ SCu300A Intrauterine Device in Comparison to TCu380 IUD Intra-uterine Contraceptive Device
Brief Title: Multivariate Assessment of the IUB Intrauterine Device Compared With a T380A IUD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ocon Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AOS-C2000
Record Dates: First submitted 2013-12-19; First posted 2014-01-14 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: To Assess the Safety, Effectiveness and User Experience of the Scu 300A IUB
Keywords: IUB

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCu300A IUB (Experimental)
  Interventions: Device: SCu300A IUB intrauterine device
- T380A copper IUD (Active Comparator)
  Interventions: Device: T380A IUD

INTERVENTIONS:
Device: SCu300A IUB intrauterine device — Spherical copper IUD
  Arms: SCu300A IUB
Device: T380A IUD — T-shaped copper IUD
  Arms: T380A copper IUD

SUMMARY:
The novel SCu300A IUB™ (hereafter IUB™) will be evaluated for safety and effectiveness in comparison with a market approved standard T shaped IUD containing 380sq.mm. of copper.

The Primary Endpoints for comparison are based on the objective and subjective parameters.

The objective parameters are pregnancy rate, perforation, expulsion and mal -position rates, changes in the endometrial thickness, rate of complications such as infection and anemia and discontinuation rates after 2 years.

The subjective parameters including Quality of Life (QoL) are: pain during insertion, menstrual characteristics and pain, bleeding in correlation to the bleeding pattern prior to insertion.

The Secondary Endpoints are physician opinion (ease of use in insertion and removal) and subject satisfaction.

ELIGIBILITY:
Inclusion criteria:

* Adult females aged 18-45
* Free and willing to fully comply with treatment process
* Healthy women seeking LARC
* Married or in a steady relationship (at least 1 year)
* Blood hemoglobin >11.5gr/dL
* Signed informed consent form
* If took COCP at least had one cycle after use of OC

Exclusion criteria:

* Use IUB/IUD as an emergency contraception
* A previously placed IUD that has not been removed
* Pregnancy or suspicion of pregnancy
* Immediately post-abortion or post-partum - unless had at least one free cycle
* Use of other contraception method (condom for either male or female, oral contraceptives, diaphragms, spermicides, hormonal patches, injections or ring, cervical cap)
* History of pelvic inflammatory disease, recent or remote.
* Postpartum endometritis or postabortal endometritis in the past 3 month
* Mucupurulent cervicitis
* Endometrial thickness more than 12 mm on insertion date
* Known anemia (except thalassemia, sickle cell, chronic anemia)
* Severe Mennorrhagia or severe Dysmenorrhea
* History of previous IUD complications
* Dysfunctional uterine bleeding
* Undiagnosed uterine bleeding
* Malignancy or suspected malignant disease of female inner or outer genitalia
* Distortions of the uterine cavity by uterine fibroids or known anatomical abnormalities
* Known intolerance or allergy to nitinol or copper and/or copper IUDs - Wilson's disease.
* Medication that may interfere with the subject's ability to complete the protocol
* Use of injectable contraception in the previous year
* Any other significant disease or condition that could interfere with the subject's ability to complete the protocol
* A history of alcohol or drug abuse
* Known infection with human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C
* Pregnancy or pregnancy planned during the year
* Enrollment (less than 30 days after completing another study) in or planned to be enrolled in another study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 366 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 24 months
Safety issues | 24 months
  Perforations, expulsions, mal-position etc
Discontinuation rate | 24 months
Patient experience | 24 months
  Recording of menstrual cramping, pain and bleeding irregularities during the trial period

SECONDARY OUTCOMES:
Physician opinion | 24 months
  Ease of use in insertion and removal

CONTACTS AND LOCATIONS:
Locations (2):
- Sofia, Bulgaria
- Spitalul Clinic "Nicolae Malaxa", Sectia Obstetri-ca-Ginecologie, Bucharest, Romania